CLINICAL TRIAL: NCT02947646
Title: Feasibility of BabyGentleStick- Adult Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Actuated Medical, Inc. (Industry)
Collaborators: Milton S. Hershey Medical Center (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Device Feasibility
Other Study IDs: STUDY00004892; R41HD088139 (NIH)
Record Dates: First submitted 2016-10-25; First posted 2016-10-28 (Estimated); Results first posted 2022-06-16 (Actual); Last update posted 2022-12-29 (Actual); Status verified 2022-05

CONDITIONS: Lack of Adverse Events; Reduced Pain Response

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- BabyGentleStick™ ON, then BabyGentleStick™ OFF (Experimental): Experimental intervention, then Active Comparator.
  Interventions: Device: BabyGentleStick™ ON; Device: BabyGentleStick™ OFF
- BabyGentleStick™ OFF, then BabyGentleStick™ ON (Experimental): Active Comparator, then Experimental intervention.
  Interventions: Device: BabyGentleStick™ ON; Device: BabyGentleStick™ OFF

INTERVENTIONS:
Device: BabyGentleStick™ ON — experimental intervention
Device: BabyGentleStick™ OFF — active comparator

SUMMARY:
This is a pilot, randomized, safety and efficacy study of an investigational device (i.e. BabyGentleStick™; BGS, Actuated Medical, Inc). The primary study objectives are to obtain subject feedback, assess device performance; and ascertain potential harm in healthy adult volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult volunteers 18-29 years of age.
* Fluent in written and spoken English
* Sex: male or female

Exclusion Criteria:

* Pregnant women
* Cognitive impairment
* Prisoner
* Individuals with known hematologic conditions or bleeding disorders
* Individuals with immune disorders where a finger lance puts them at risk for infection.

Ages: 18 Years to 29 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2016-11; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Clement, Ph.D., Principal Investigator — Actuated Medical, Inc.; Kim K Doheny, Ph.D., Principal Investigator — The Pennsylvania State University College of Medicine
Locations (1):
- Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- BabyGentleStick™ ON, Then BabyGentleStick™ OFF: Experimental intervention first (5 minutes), followed by Active Comparator (5 minutes).
- BabyGentleStick™ OFF, Then BabyGentleStick™ ON: Active Comparator first (5 minutes), then Experimental intervention (5 minutes).
Period: Overall Study
Arm/Group | BabyGentleStick™ ON, Then BabyGentleStick™ OFF | BabyGentleStick™ OFF, Then BabyGentleStick™ ON
Started | 10 | 10
Completed | 10 | 9
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- BabyGentleStick™ ON, Then BabyGentleStick™ OFF: Experimental intervention followed by Active Comparator.
- BabyGentleStick™ OFF, Then BabyGentleStick™ ON: Active Comparator followed by Experimental intervention.
- Total: Total of all reporting groups
Arm/Group | BabyGentleStick™ ON, Then BabyGentleStick™ OFF | BabyGentleStick™ OFF, Then BabyGentleStick™ ON | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 10 | 20
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 8 | 8 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | NA — race/ethnicity data not collected | NA — race/ethnicity data not collected | NA — Total not calculated because data are not available (NA) in one or more arms.
  Not Hispanic or Latino | NA — race/ethnicity data not collected | NA — race/ethnicity data not collected | NA — Total not calculated because data are not available (NA) in one or more arms.
  Unknown or Not Reported | NA — race/ethnicity data not collected | NA — race/ethnicity data not collected | NA — Total not calculated because data are not available (NA) in one or more arms.
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: Number of Adverse Events
Description: Subjects will receive a follow-up phone call 24 hours post-intervention to monitor adverse events.
Time Frame: 24 hours after the intervention is received for each subject
Measure: Number; unit: events
Groups:
- BabyGentleStick™ ON: Experimental intervention, whether it was performed first or was performed after Active Comparator
- BabyGentleStick™ OFF: Active Comparator, whether it was performed first or was performed after Experimental intervention
Arm/Group | BabyGentleStick™ ON | BabyGentleStick™ OFF
Number analyzed (Participants) | 19 | 20
events | 0 | 1

2. Secondary Outcome: Reduced Pain Response
Description: Relative Likert pain scale from 1 to 10, with 0 being no pain and 10 being extreme pain.
Time Frame: 5 minutes
Measure: Mean (Standard Deviation); unit: score on a Likert scale
Groups:
- BabyGentleStick™ ON: Experimental intervention, whether it was performed first or was performed after the Active Comparator.
- BabyGentleStick™ OFF: Active Comparator, whether it was performed first or was performed after the Experimental intervention.
Arm/Group | BabyGentleStick™ ON | BabyGentleStick™ OFF
Number analyzed (Participants) | 19 | 20
score on a Likert scale | 1.74 (1.45) | 1.80 (1.24)

ADVERSE EVENTS:
Time Frame: 1 day
Groups:
- BabyGentleStick™ ON: Experimental intervention to be compared to the Active Comparator.
  BabyGentleStick™ ON
- BabyGentleStick™ OFF: Active Comparator intervention to be compared to the Experimental interventional.
  BabyGentleStick™ OFF
Arm/Group | BabyGentleStick™ ON | BabyGentleStick™ OFF
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/20
Other Adverse Events (participants affected / at risk) | 0/19 | 1/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BabyGentleStick™ ON (N=19) | BabyGentleStick™ OFF (N=20)
Unexpected bleeding (Blood and lymphatic system disorders) | 0 | 1 — Unexpected bleeding with first lancet puncture (vibration off). Required pressure to site for >12 min to stop bleeding. PI elected to stop study for this enrollee and not perform procedure with vibration on.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No